CLINICAL TRIAL: NCT03982628
Title: Rates of Sarcopenia Development Using Abdominal CT Imaging in the Critically Ill With Sepsis Compared to the Critically Ill With Trauma
Brief Title: ICU Sarcopenia Rates by Abdominal CT: Sepsis vs. Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB19-0595
Record Dates: First submitted 2019-05-14; First posted 2019-06-11 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2019-05

CONDITIONS: Sarcopenia; Critical Illness; Sepsis; Trauma
MeSH Terms: conditions — Sarcopenia; Critical Illness; Sepsis; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Adults admitted to a mixed medical/surgical ICU for sepsis with at least two abdominal CT imaging studies separated by at least 24 hours, ordered as part of their routine clinical care.
  Interventions: Diagnostic Test: Abdominal CT imaging
- Trauma: Adults admitted to a mixed medical/surgical ICU for trauma (without sepsis) with at least two abdominal CT imaging studies separated by at least 24 hours, ordered as part of their routine clinical care.
  Interventions: Diagnostic Test: Abdominal CT imaging

INTERVENTIONS:
Diagnostic Test: Abdominal CT imaging — Routine abdominal CT imaging

SUMMARY:
Using abdominal computed tomography (CT) imaging, the investigators will estimate total body muscle mass at two time points in Intensive Care Unit (ICU) by assessing cross-sectional muscle areas at the L3 vertebral body level. This allows for a determination of the rate of sarcopenia development in the ICU.

With this information, the investigators propose to test if the rates of the development of sarcopenia differ in critically ill subjects with sepsis compared to a reference group of critically ill subjects with trauma (without sepsis).

DETAILED DESCRIPTION:
The investigators propose to compare rates of development of sarcopenia in critically ill, septic subjects with a reference cohort of critically ill, trauma subjects who are not septic. The null hypothesis is that the rates of muscle loss in subjects with sepsis (a condition associated with high levels of inflammation) are comparable with the rates of muscle loss in subjects without sepsis. As secondary outcomes, the investigators will evaluate whether rates of muscle loss correlate with clinical assessments in the ICU (body mass index, frailty score, illness severity score), with clinical course through the hospital (ICU length of stay (LOS), duration of mechanical ventilation, hospital LOS, ICU readmissions, hospital readmissions), and with outcomes (discharge destination, ICU mortality, hospital mortality and six-month mortality).

To answer this question, the investigators propose to retrospectively analyze existing abdominal CT imaging of subjects treated in the ICU. Muscle mass estimations will be performed by determining skeletal muscle cross-sectional area for muscles at the level of the L3 vertebra using previously validated techniques. The CT images will have been gathered as part of routine care for subjects admitted to a mixed medical-surgical ICU. These data will be correlated with anonymized clinical and demographic information. Study participants will be grouped into two cohorts - subjects admitted to the ICU for sepsis, and subjects admitted to the ICU for trauma. People who experience both trauma and sepsis will be excluded. Only subjects with at least 2 or more abdominal CT imaging event will be included.

Results from this study will be assessed using a generalized linear model to determine if the two groups are different. From earlier studies, the investigators estimate that 73 subjects will be required in each group to detect between-group differences for the primary outcome.

The results of this study will add to the general understanding of the rates of muscle loss in a critical care setting for subjects admitted to ICU with sepsis, as compared to subjects with trauma. Secondary outcome information will be presented descriptively to show sarcopenia rates for the two cohorts, in the context of select clinical, demographic and administrative variables.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU with sepsis or trauma
* Two abdominal CT imaging tests (separated by at least 24 hours, within the first 3 weeks of their ICU admission) performed as part of their routine clinical care.

Exclusion Criteria:

* Children (age < 18 years)
* Repeat admission to ICU within the previous 6 months
* Medical or neurological diagnosis that may plausibly affect the muscle bulk of the muscles at the L3 vertebra body level (e.g. achondroplasia, spinal muscular atrophy, spinal cord injury, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are comparing muscle mass estimations based on previously ordered serial abdominal CT imaging. We are comparing sepsis to a reference group of trauma without sepsis. We anticipate that the sepsis group will contain subjects with abdominal sepsis primarily (as this would be a trigger for clinically testing patients with repeat abdominal CT imaging). We anticipate the the trauma cohort will consist of primarily splenic lacerations that are being monitored clinically, although this group will also likely contain patients with liver, renal, and intestinal injuries related to trauma.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of sarcopenia development | Sarcopenia assessed over their admission to ICU (to a ceiling of the first 3 weeks of ICU)
  Described as a percentage loss of muscle mass per day (%/d)

SECONDARY OUTCOMES:
Sarcopenia's correlation with clinical assessments in ICU - Body Mass Index | Sarcopenia assessed over the first 3 weeks of admission to ICU, body mass index calculated from clinical assessment on the day of CT imaging
  Association of sarcopenia (%/d) with body mass index (kg/m^2)
Sarcopenia's correlation with clinical assessments in ICU - Clinical Frailty Score | Sarcopenia assessed over the first 3 weeks of admission to ICU, clinical frailty scale assessed at admission to ICU
  Association of sarcopenia (%/d) with clinical frailty score (a descriptive integer ranging from 1, meaning "Very Fit", to 9, meaning "Terminally Ill") as assessed by the subject's admitting ICU physician
Sarcopenia's correlation with clinical assessments in ICU - Sequential Organ Failure Assessment (SOFA) score | Sarcopenia assessed over the first 3 weeks of admission to ICU, SOFA scores calculated from clinical variables on the first day of admission to the ICU
  Association of sarcopenia (%/d) with illness severity as described by the SOFA score (an integer between 0 and 24 where the scores are determined by the health of 6 organ systems. Higher SOFA scores indicate higher chances of mortality)
Sarcopenia's correlation with clinical course - ICU length of stay | Sarcopenia assessed over the first 3 weeks of admission to ICU, ICU LOS calculated from ICU admission to discharge (to a ceiling of 180 days)
  Association of sarcopenia (%/d) with ICU LOS (d)
Sarcopenia's correlation with clinical course - Hospital length of stay | Sarcopenia assessed over the first 3 weeks of admission to ICU, hospital LOS calculated from hospital admission to discharge (to a ceiling of 180 days)
  Association of sarcopenia (%/d) with hospital LOS (d)
Sarcopenia's correlation with clinical course - Duration of mechanical ventilation | Sarcopenia assessed over the first 3 weeks of admission to ICU, duration of mechanical ventilation calculated from initiation of mechanical ventilation within the hospital stay of interest to ventilator weaning (to a ceiling of 180 days)
  Association of sarcopenia (%/d) with duration of mechanical ventilation (d)
Sarcopenia's correlation with subject outcomes - ICU mortality | Sarcopenia assessed over the first 3 weeks of admission to ICU, ICU mortality calculated as the percentage of subjects who do not survive to ICU discharge (to a ceiling of 180 days)
  Association of sarcopenia (%/d) with percentage survival to ICU discharge (%)
Sarcopenia's correlation with subject outcomes - Hospital mortality | Sarcopenia assessed over the first 3 weeks of admission to ICU, hospital mortality calculated as the percentage of subjects who do not survive to hospital discharge (to a ceiling of 180 days)
  Association of sarcopenia (%/d) with percentage survival to hospital discharge (%)
Sarcopenia's correlation with subject outcomes - Change in living setting | Sarcopenia assessed over the first 3 weeks of admission to ICU, change in living setting calculated as the percentage of subjects discharge to an alternate living setting at hospital discharge (to a ceiling of 180 days)
  Association of sarcopenia (%/d) with percentage of subjects discharged from hospital to their pre-critical illness living setting (%)
Sarcopenia's correlation with subject outcomes - Six-month mortality | Sarcopenia assessed over the first 3 weeks of admission to ICU, Six-month mortality calculated as the percentage of subjects deceased at 180 days after ICU admission
  Association of sarcopenia (%/d) with percentage of subjects alive 180 days after their ICU admission (%)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Grant, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No